CLINICAL TRIAL: NCT03078439
Title: Epidemiologic Study on Small-for-gestational-age Children (EPIPAGE2 Cohort Study) - Follow up at Five and a Half Years
Brief Title: EPIPAGE2 Cohort Study Follow up at Five and a Half Years
Acronym: EPIPAGE2
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C15-95; IDRCB (Registry Identifier: 2016-A00333-48)
Record Dates: First submitted 2016-11-08; First posted 2017-03-13 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2021-08

CONDITIONS: Very Preterm Birth
Keywords: very preterm birth; developmental disorders; health problems; prospective population-based cohort
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — DNA from saliva samples collected from 5 years and a half children
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Medical and neuropsychological assessments — Assessment of health status and development will be performed in specific centers at 5 and a half years. This check-up includes a complete medical examination to look for visual, hearing, motor impairment and health problems, and psychological tests using standardized tools (WPPSI IV ((Wechsler Preschool and Primary Scales Intelligence)) and NEPSY 2 tests) to assess cognitive development of very preterm children.
  A parental questionnaire will be fulfilled to investigate family's social conditions, maternal health, autism spectrum disorders (Social Communication Questionnaire), the child's quality of life and behavioral development (Strengths and Difficulties Questionnaire).

SUMMARY:
Epipage 2 (epidemiologic study on small-for-gestational-age children) is a nationwide study implemented to improve our knowledge of the outcome of preterm children in France. This study was launched on March 28, 2011 and includes three groups of preterm children, all born before 35 weeks: extremely preterm infants (born between 22 and 26 completed weeks of gestation), very preterm children (born between 27 and 31 completed weeks) and moderately preterm children (born between 32 and 34 completed weeks).

These children are being studied from their birth up to the age of 12 years. At birth, data on maternal and infants' characteristics were collected from medical records. At one and two years, questionnaires sent to families and to physicians (at two years only) allowed to collect data about the children's life and health.

At five and a half years, medical and psychological assessments are specifically implemented for the study in order to evaluate motor and cognitive disorders in this population.

ELIGIBILITY:
Inclusion Criteria:

* initially included in EPIPAGE 2 cohort or complementary studies or Elfe cohort study
* family agreement to participate to cohort follow up
* informed consent form signed by both parents
* affiliated to social security system

Exclusion Criteria:

* parental refusal
* not affiliated to any social security system

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm children included at birth in the EPIPAGE 2 cohort or in complementary studies whose famillies agree to participate to EPIPAGE 2 follow up (4600 children) + 600 children born at term and participating to the Elfe cohort (French longitudinal study of children)
Sampling Method: Probability Sample
Enrollment: 3404 (Actual)
Dates: Start 2016-09-02 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2018-01-08 (Actual)

PRIMARY OUTCOMES:
Health disorders assessed by medical exam | 5 years 5 months- 5 years 11 months
  According to gestational age at birth
Motor disorders assessed by medical exam | 5 years 5 months- 5 years 11 months
  According to gestational age at birth
Cognitive disorders assessed by psychological testing | 5 years 5 months- 5 years 11 months
  According to gestational age at birth
Behavioural disorders by psychological testing | 5 years 5 months- 5 years 11 months
  According to gestational age at birth

SECONDARY OUTCOMES:
Changes in medical practices collected by questionnaire | 5 years 5 months- 5 years 11 months
Changes in organization of care collected by questionnaire | 5 years 5 months- 5 years 11 months
Set up a DNA Biobank by saliva samples collection | 5 years 5 months- 5 years 11 months

CONTACTS AND LOCATIONS:
Locations (98):
- France (92):
  - Centre Hopsitalier d'Agen, Agen
  - CAMSP Albi, Albi
  - CHU Amiens, Amiens
  - CHU d'Angers, Angers
  - CH d'Arras, Arras
  - CAMSP Auch, Auch
  - Centre Hospitalier Côte Basque, Bayonne
  - CH Beauvais, Beauvais
  - CHU Jean Minjoz, Besançon
  - Centre Hospitalier de Bordeaux, Bordeaux
  - CH Bourg en Bresse, Bourg-en-Bresse
  - CHU de Brest, Brest
  - Rezo Camsp, Brioude
  - Hopital Femme, Mère, Enfant, Bron
  - CHU de Caen, Caen
  - CH Cahors, Cahors
  - CMPP de Cahors, Cahors
  - CH de Calais, Calais
  - CH de Carcassonne, Carcassonne
  - CH Castres - Hôpital du pays d'Autan, Castres
  - CH Chalon sur Saone - William Morey, Chalon-sur-Saône
  - Réseau Eclaur, Chambéry
  - CH Métropole Savoie, Chambéry
  - CAMSP de Charleville Mézières, Charleville-Mézières
  - CHU Estaing, Clermont-Ferrand
  - Centre Hospitalier de Colmar, Colmar
  - CH Compiègne, Compiègne
  - CH Alpes Leman, Contamine-sur-Arve
  - CH Sud Francilien, Corbeil
  - CH Creil, Creil
  - CAMSP de Dax, Dax
  - CHU Dijon - Hôpital du Bocage, Dijon
  - CH de Douai, Douai
  - CAMSP Espaly, Espaly-Saint-Marcel
  - SCM Maison de l'enfant, Essey-lès-Nancy
  - Hôpital d'Epinal, Épinal
  - Hôpital de Forbach, Forbach
  - CHU Grenoble / Réseau Naitre et Devenir, Grenoble
  - Centre Hospitalier de Haguenau, Haguenau
  - CH Laon, Laon
  - CHU Le Mans, Le Mans
  - CH de Lens, Lens
  - Hôpital Saint Vincent de Paul - Groupement des Hôpitaux de l'Institut Catholique de Lille, Lille
  - CHRU de Lille, Lille
  - Hôpital Mère-Enfant de Limoges, Limoges
  - CAMSP, CHU de Lorient, Lorient
  - Hopital de la Croix Rousse, Lyon
  - CHU Hôpital Nord, Marseille
  - CHU de la Conception, Marseille
  - CH de Maubeuge, Maubeuge
  - CH Mâcon, Mâcon
  - Hôpital de Mercy - CHR Metz Thionville, Metz
  - CH Annecy Genevois, Metz-Tessy
  - Centre Hospitalier de Mont de Marsan, Mont-de-Marsan
  - CAMSP "l'Escabelle" Montauban, Montauban
  - CH Montauban, Montauban
  - GHH Havre - Hôpital Jacque Monod, Montivilliers
  - CHU de Montpellier, Montpellier
  - CAMSP - CHU Saint-Eloi, Montpellier
  - Centre Hospitalier de Mulhouse, Mulhouse
  - CHRU de Nancy (Maternité), Nancy
  - CHRU de Nancy (Neuro-pédiatrie), Nancy
  - CHU de Nantes, Nantes
  - CHU Hôpital l'Archet, Nice
  - CHU de Nimes - Hôpital Caremeau, Nîmes
  - CHR Orléans, Orléans
  - Hôpital Armand Trousseau, Paris
  - CIC Necker, Paris
  - Centre Hospitalier de Pau, Pau
  - CHG de Perpignan (CAMSP), Perpignan
  - CAMSP de Périgueux, Périgueux
  - CHU de Reims / CAMSP, Reims
  - CAMSP, CHU de Rennes, Rennes
  - CH Rodez - Jacques Puel, Rodez
  - CH de Roubaix, Roubaix
  - CHU de Rouen - Pavillon Mère et enfant, Rouen
  - CAMSP de Saint Brieuc, Saint-Brieuc
  - CHU Sud Réunion, Saint-Pierre
  - CHU St Etienne / Réseau HELENA, Saint-Priest-en-Jarez
  - CH Saint Quentin, Saint-Quentin
  - Centre Hospitalier Hautepierre, Strasbourg
  - CH de Bigorre, Tarbes
  - CAMSP Thionville, Thionville
  - Hôpital Bel Air Thionville - CHR Metz Thionville, Thionville
  - CHU de Toulouse - Hôpital des enfants, Toulouse
  - Clinique Ambroise Paré, Toulouse
  - CHRU de Tours -Hôpital Clocheville, Tours
  - CAMSP de Troyes, Troyes
  - CH Valence, Valence
  - CH de Valenciennes, Valenciennes
  - CH de Vannes, Vannes
  - CH Villefranche sur Saone, Villefranche-sur-Saône
- French Guiana (2):
  - CH Andrée Rosemon, Cayenne
  - CH de l'Ouest Guyanais, Saint-Laurent-du-Maroni
- Guadeloupe (2):
  - CAMSP Basse-Terre, Basse-Terre
  - CHU Pointre à Pitre, Les Abymes
- Reunion (2):
  - CAMSP Nord-ASFA Sainte Clotilde, Saint-Denis
  - CHU Felix Guyon, Saint-Denis

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guellec I, Brunet A, Lapillonne A, Taine M, Torchin H, Favrais G, Gascoin G, Simon L, Heude B, Scherdel P, Kayem G, Delorme P, Jarreau PH, Ancel PY. Birth weight and head circumference discordance and outcome in preterms: results from the EPIPAGE-2 cohort. Arch Dis Child. 2024 May 17;109(6):503-509. doi: 10.1136/archdischild-2023-326336. PMID 38408861
- See also: Epipage 2 website — http://epipage2.inserm.fr/